CLINICAL TRIAL: NCT02411942
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study Comparing Adapalene Gel 0.3% to Differin® (Adapalene Gel 0.3%) and Both Active Treatments to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Adapalene Gel 0.3% to Differin® and Both to a Placebo Control in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADPG 1410
Record Dates: First submitted 2015-04-04; First posted 2015-04-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adapalene Gel 0.3% (Experimental): Adapalene Gel 0.3% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Adapalene Gel 0.3%
- Differin® (Active Comparator): Differin® (adapalene gel 0.3%) (Galderma Laboratories, LP, US)
  Interventions: Drug: Differin®
- Placebo (Placebo Comparator): Placebo (vehicle of the test product) (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene Gel 0.3% — Adapalene Gel 0.3% applied to the entire face once daily for 84 consecutive days
  Other Names: Adapalene
  Arms: Adapalene Gel 0.3%
Drug: Differin® — Differin® applied to the entire face once daily for 84 consecutive days
  Other Names: Adapalene
  Arms: Differin®
Drug: Placebo — Placebo (vehicle of the test product) applied to the entire face once daily for 84 consecutive days
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the therapeutic equivalence and safety of Adapalene Gel 0.3% and Differin® (adapalene gel 0.3%).

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the therapeutic equivalence and safety of Adapalene Gel 0.3% and Differin® (adapalene gel 0.3%) in the treatment of acne vulgaris and to demonstrate the superiority of the efficacy of the test and reference products over the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects aged 18 years and older must have provided written consent. Subjects aged 12 to 17 years must have provided written assent accompanied by written consent from their legally acceptable representative. All subjects or their legally acceptable representatives must sign Health Insurance Portability and Accountability Act authorization.
* Must have a minimum of ≥ 25 non-inflammatory lesions and ≥ 20 inflammatory lesions and ≤ 2 nodulocystic lesions at baseline on the face.
* Must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Have a history of hypersensitivity or allergy to adapalene, retinoids and/or any of the study medication ingredients.
* Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 753 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Change in non-inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts

SECONDARY OUTCOMES:
Clinical response of success | Week 12
  The proportion of subjects with a clinical response of success at week 12, success defined as an Investigator's Global Assessment score that is at least two grades less than the baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/